CLINICAL TRIAL: NCT06927427
Title: Evaluation of Swallowing Impairment After Tonsillectomy: A Cohort Study
Brief Title: Evaluation of Swallowing Impairment After Tonsillectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: FMASU MS75/2024
Record Dates: First submitted 2025-04-04; First posted 2025-04-15 (Actual); Last update posted 2025-04-15 (Actual); Status verified 2024-02

CONDITIONS: Swallowing Impairment After Tonsillectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Post tonsillectomy group (Other)
  Interventions: Procedure: fiberoptic endoscopic evaluation of swallowing (FEES)

INTERVENTIONS:
Procedure: fiberoptic endoscopic evaluation of swallowing (FEES) — Using flexible endoscopy, the patient will be given a colored thin fluid to keep in their mouth and then swallow following the instructions of the examiner, then the examination will be repeated using semisolids (1 teaspoon of yogurt) and using solids (piece of bread). The evaluation of swallowing will involve four items: early spill of food (delayed triggering), aspiration, penetration, and retention (residue). And the results will be recorded.

SUMMARY:
the investigator will evaluate the swallowing pattern of the patients pre-operative and will follow them up at day 15 after tonsillectomy by using Careful history taking and Fiberoptic endoscopic evaluation of swallowing (FEES).

DETAILED DESCRIPTION:
All patients will be evaluated pre-operative by history taking using the Arabic version of Eating Assessment Tool (EAT-10) questionnaire and will be examined by Fiberoptic endoscopic evaluation of swallowing (FEES). All patients will be operated by the same surgical technique. Patients will be directed to return back on the 15th day post-operative after tonsillectomy and they will be subjected to history taking using the Arabic version of Eating Assessment Tool (EAT-10) questionnaire and they will be examined by Fiberoptic endoscopic evaluation of swallowing (FEES).

1. Careful history taking The history of the patients will be taken using the Arabic version of the Eating Assessment Tool (EAT-10) questionnaire. The patient will rate the problem on a scale of 0 to 4 (0 means no problem; 4 means severe problem). A score of 3 or more on the EAT-10 is considered dysphagia.
2. Fiberoptic endoscopic evaluation of swallowing (FEES). Using flexible endoscopy (the flexible nasopharyngeal video-fiberscope Henke-Sass-Wolf, 4.3mm in diameter connected to Lemke video camera). The patient will be given a colored thin fluid to keep in their mouth and then swallow following the instructions of the examiner, then the examination will be repeated using semisolids (1 teaspoon of yogurt) and using solids (piece of bread). The evaluation of swallowing will involve four items: early spill of food (delayed triggering), aspiration, penetration, and retention (residue). And the results will be recorded.

ELIGIBILITY:
Inclusion Criteria:

1. Patients undergoing tonsillectomy.
2. Age group (from 7-18 years).
3. Patients of either gender.

Exclusion Criteria:

1. Patients younger than 7 years or older than 18 years.
2. Patients with neurological diseases and genetic syndromes.
3. Patients with history of swallowing disorders prior to tonsillectomy.

Ages: 7 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 20 (Actual)
Dates: Start 2024-06-01 (Actual); Primary Completion 2024-12-01 (Actual); Study Completion 2025-01-01 (Actual)

PRIMARY OUTCOMES:
evaluation of swallowing impairment after tonsillectomy | 15 days after tonsillectomy
  To evaluate the swallowing process in children after tonsillectomy and detect the occurance of dysphagia. using the Arabic version of the Eating Assessment Tool (EAT-10) questionnaire, the patient will rate the problem on a scale of 0 to 4 (0 means no problem; 4 means severe problem). A score of 3 or more on the EAT-10 is considered dysphagia. And Fiberoptic endoscopic evaluation of swallowing (FEES), the evaluation of swallowing will involve four items: early spill of food (delayed triggering), aspiration, penetration, and residue.

CONTACTS AND LOCATIONS:
Overall Officials: Alaa A Mansour, MBBCH, Principal Investigator — OtoRhinoLaryngology, head and neck surgery resident, Ain Shams University
Locations (1):
- Ain Shams University, Cairo, Cairo Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Yes
all data will be shared once study is completed
Supporting Information: Study Protocol, SAP, ICF
Time Frame: once study is completed
Access Criteria: free